CLINICAL TRIAL: NCT05620160
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study of RAY1216 Tablets in Patients With Mild to Moderate SARS-CoV-2 Infection
Brief Title: Study of RAY1216 Tablets Compared With Placebo in Patients With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAY1216-22-02
Record Dates: First submitted 2022-11-04; First posted 2022-11-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Mild to Moderate COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAY1216 (Experimental): Participants received 400mg RAY1216 tablet orally three times daily for 5 days.
  Interventions: Drug: RAY1216
- Placebo (Placebo Comparator): Participants received 400mg placebo orally three times daily for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAY1216 — RAY1216（tablet）
  Arms: RAY1216
Drug: Placebo — placebo （tablet）
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled clinical trial to assess the efficacy and safety of RAY1216 tablets in the treatment of mild to moderate SARS-CoV-2 infection. The total study duration is up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who provide written informed consent before the trial, and fully understand the trial content, process and possible adverse reactions.
2. Participants who are willing and able to comply with the protocol for treatment plan, virological testing, laboratory testing and other study procedures.
3. Male or female participants aged 18-75 (including 18 and 75 years old).
4. Confirmed SARS-CoV-2 infection 120 hours prior to randomization.
5. Initial onset of COVID-19 symptoms/signs within 48 hours before randomization.
6. Fertile participants must agree to take effective contraceptive measures.

Exclusion Criteria:

1. Patients with severe or critical COVID-19 who currently require hospitalization, or patients who are expected to develop into severe or critical disease and require hospitalization within 48h after randomization.
2. Difficulty swallowing or a history of gastrointestinal diseases that seriously affect drug absorption.
3. Active liver disease, or obvious abnormal liver function (ALT or AST ≥ 3ULN, or total bilirubin ≥ 2ULN).
4. WBC >1ULN, or NEU <0.5ⅹ109/L.
5. Receiving dialysis or have known moderate to severe renal impairment (eGFR<60mL/min/1.73m2).
6. Other suspected or confirmed systemic infections.
7. Current or expected use of strong CYP3A4 inducers, inhibitors or medications that are highly dependent on CYP3A4 or CYP2C19 for clearance.
8. Prior or anticipated receipt of any vaccine within 28 days prior to enrollment and during study period.
9. Use of antivirals against SARS-CoV-2 within 7 days prior to enrollment.
10. Weight≤40kg.
11. Pregnant, lactating women or those with a positive pregnancy test (sterilized or postmenopausal women may not have a pregnancy test).
12. Previous administration with any investigational drug within 3 months before the study drug administration.
13. Participants who are judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1359 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Time to sustained clinical recovery of 11 COVID-19 symptoms | Day 1 through Day 29
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 for three consecutive days.

SECONDARY OUTCOMES:
Proportion of participants who experience hospitalization or death cause by progression to severe disease | Day 1 through Day 29
Proportion of participants who experience death from any cause | Day 1 through Day 29
Proportion of participants who experience COVID-19 related hospitalization or death from any cause | Day 1 through Day 29
SARS-CoV-2 viral shedding time in nasopharyngeal swabs | baseline, Day 4, Day 6, Day 10, Day 15
Change of viral load compared to the baseline | baseline, Day 4, Day 6, Day 10, Day 15
Proportion of participants who are negative for SARS-CoV-2 nucleic acid test | baseline, Day 4, Day 6, Day 10, Day 15
Time to clinical sustained remission | Day 1 through Day 29
Proportion of participants in clinical recovery/remission | Day 1 through Day 29
Time to sustained clinical recovery of 10 COVID-19 symptoms except cough | Day 1 through Day 29
Time to sustained clinical recovery of COVID-19 respiratory and systemic symptoms | Day 1 through Day 29
Time to sustained clinical recovery of each COVID-19 targeted symptoms | Day 1 through Day 29
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 through Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhan Y, Lin Z, Liang J, Sun R, Li Y, Lin B, Ge F, Lin L, Lu H, Su L, Xiang T, Pan H, Huang C, Deng Y, Wang F, Xu R, Chen D, Zhang P, Tong J, Wang X, Meng Q, Zheng Z, Ou S, Guo X, Yao H, Yu T, Li W, Zhang Y, Jiang M, Fang Z, Song Y, Chen R, Luo J, Kang C, Liang S, Li H; other Collaborative Institutes; Zheng J, Zhong N, Yang Z. Leritrelvir for the treatment of mild or moderate COVID-19 without co-administered ritonavir: a multicentre randomised, double-blind, placebo-controlled phase 3 trial. EClinicalMedicine. 2023 Dec 14;67:102359. doi: 10.1016/j.eclinm.2023.102359. eCollection 2024 Jan. PMID 38188690